CLINICAL TRIAL: NCT03124927
Title: Accuracy of Methemoglobin Measurement for Rainbow DCI Sensors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR-17413-REDF0003
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Results first posted 2017-06-12 (Actual); Last update posted 2017-06-12 (Actual); Status verified 2017-05

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test Group (Experimental): All subjects are enrolled into the test group and all subjects receive DCI pulse oximeter sensor.
  Interventions: Device: DCI pulse oximeter sensor

INTERVENTIONS:
Device: DCI pulse oximeter sensor

SUMMARY:
In this study, the level of methemoglobin (HbMet) will be increased in a controlled manner by administering sodium nitrite intravenously in healthy volunteers. The accuracy of a noninvasive HbMet measurement by a DCI pulse oximeter sensor will be assessed by comparison to blood measurements from a laboratory analyzer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must understand and consent to be in the study
2. American Society of Anesthesiology Class I (Healthy subjects without any systemic disease at all).

Exclusion Criteria:

1. Subjects who have any systemic disease at all.
2. Subjects who do not understand the study and the risks involved.
3. Current smokers.
4. Subjects who are pregnant.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-04-23 (Actual); Primary Completion 2008-08-08 (Actual); Study Completion 2008-08-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - University of California, San Francisco, San Francisco, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test Group
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Test Group
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Sensor by Arms Calculation
Description: Accuracy will be determined by comparing the noninvasive blood methemoglobin measurement of the pulse oximeter to that obtained from a blood sample and calculating the arithmetic root mean square (Arms) error value.
Time Frame: 5 hours
Measure: Number; unit: percentage
Arm/Group | Test Group
Number analyzed (Participants) | 25
percentage | 0.87

ADVERSE EVENTS:
Arm/Group | Test Group
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less